CLINICAL TRIAL: NCT01137851
Title: Effect of Patient Cost Sharing on Treatment Discontinuation Among Rheumatoid Arthritis Patients Treated With Biologic Disease Modifying Antirheumatic Drug (DMARD) Therapies
Brief Title: Effect of Patient Cost Sharing on Treatment Discontinuation Among Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: IM101-256
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New to bDMARD: New to bDMARD RA patients with high and low cost share who continue or discontinue treatment

SUMMARY:
The purpose of this study is to assess the impact of patient cost sharing on treatment discontinuation of biologic agents in patients with Rheumatoid Arthritis (RA)

ELIGIBILITY:
Patients diagnosed with Rheumatoid Arthritis (RA) who newly initiated a biologic DMARD (bDMARD) during a study timeframe of 1/01/06 to 3/31/09.

Inclusion Criteria:

* 18 to 64 years of age at index date
* Diagnosis of RA during the study period (ICD-9CM 714.xx)
* Evidence of at least one biologic DMARD of interest during the study timeframe
* Continuous enrollment during the study timeframe
* Both medical and pharmacy benefits
* No evidence of a claim for a bDMARD in the 6-month pre-period

Exclusion Criteria:

* Patients are excluded if they have a diagnosis of psoriasis, psoriatic arthritis, ankylosing spondylitis, Crohn's disease, or ulcerative colitis at any time during the study timeframe; have a claim for Rituxan, IV etanercept, or IV adalimumab; or have Medicare or Medicaid during the study timeframe

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial health plan members
Sampling Method: Probability Sample
Enrollment: 3940 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Effect of patient cost share on discontinuation | Assessed from first prescription date and followed for 1-year

SECONDARY OUTCOMES:
RA-related healthcare utilization and costs | Pre-index: 6-month period prior to the index drug date
All-cause healthcare utilization and costs | Pre-index: 6-month period prior to the index drug date
RA-related healthcare utilization and costs | Post-period: Index date+365 days
All-cause healthcare utilization and costs | Post-period: Index date+365 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm